CLINICAL TRIAL: NCT06588686
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Trial Evaluating the Efficacy and Safety of 2 Doses of Buloxibutid Over 52 Weeks in People With Idiopathic Pulmonary Fibrosis.
Brief Title: A Trial to Evaluate Efficacy and Safety of Buloxibutid in People With Idiopathic Pulmonary Fibrosis.
Acronym: ASPIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Collaborators: Population Services International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-C21-011
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Angiotensin, IPF, angiotensin II receptor 2, buloxibutid
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — compound 21

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Buloxibutid 100 mg BID (Experimental): For 52 weeks.
  Interventions: Drug: Buloxibutid
- Buloxibutid 50 mg BID (Experimental): For 52 weeks.
  Interventions: Drug: Buloxibutid
- Placebo BID (Placebo Comparator): For 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buloxibutid — Buloxibutid
  Other Names: C21
  Arms: Buloxibutid 100 mg BID; Buloxibutid 50 mg BID
Drug: Placebo — Placebo
  Arms: Placebo BID

SUMMARY:
The ASPIRE trial is a 52 week randomized, double-blind, placebo-controlled, parallel-group, multicenter trial in which the efficacy, safety, and pharmacokinetics of orally administered buloxibutid, either on top of stable IPF therapy or as monotherapy, are assessed in participants with IPF.

Trial website: www.aspire-ipf.com

DETAILED DESCRIPTION:
Buloxibutid is an oral angiotensin II type 2 (AT2) receptor agonist and has been shown to improve lung function in IPF over 36 weeks.

Buloxibutid agonizes the AT2 receptor on alveolar epithelial type 2 cells (AEC2s), which are believed to play a central role in the disease. Buloxibutid has been demonstrated preclinically to improve AEC2 viability, alveolar integrity via surfactant secretion and epithelial repair via replenishment of gas exchange alveolar epithelial type 1 cells (AEC1s). This leads to decreasing downstream profibrotic signaling, enhancing resolution of existing fibrotic tissue via upregulation of collagenase matrix metalloproteinases, and addressing vascular disfunction associated with the disease.

The trial will include participants who are on stable licensed IPF therapy or who are currently not treated with a licensed IPF therapy. The latter group will include participants intolerant or not responsive to licensed IPF therapies, participants ineligible to receive these therapies, and participants who have voluntarily declined to receive a licensed IPF therapy after being fully informed of the potential benefits and risks of such therapy. Due to the potential risk of drug-drug interactions (DDIs), concomitant treatment with pirfenidone is not allowed in this trial. Participants who are not on antifibrotic therapy at study start may initiate such treatment during the study.

The trial is planned to enroll 360 participants, 120 participants on oral buloxibutid 100 mg BID, 120 participants on oral buloxibutid 50 mg BID, and 120 participants on oral placebo BID for 52 weeks. The treatment will be blinded and treatment allocation will be randomized.

The primary measurement will be based on spirometry, measuring the forced vital capacity (FVC).

The trial consists of 3 consecutive periods: a screening period of up to 6 weeks, a 52-week treatment period, and a follow-up period of 2-4 weeks after the 52-week visit. The study procedures have been planned with focus on optimizing patient convenience while allowing a safe conduct and strict scientific rigor.

Trial website: www.aspire-ipf.com

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 40 years at the time of signing the informed consent.
2. Diagnosed with IPF within 7 years prior to visit 1, as per applicable ATS/ERS/JRS/ALAT guidelines at the time of diagnosis.
3. HRCT scan within 36 months prior to visit 1 with central reading confirming either a or b, and c

   1. A pattern consistent with usual interstitial pneumonia (UIP) according to ATS/ERS/JRS/ALAT 2022 guideline (Raghu et al., 2022) UIP or probable UIP.
   2. A pattern indeterminate for UIP according to ATS/ERS/JRS/ALAT 2022 guidelines (Raghu et al., 2022) and a historical biopsy (surgical lung biopsy or transbronchial lung cryobiopsy) consistent with IPF.
   3. Extent of fibrosis > extent of emphysema.
4. FVC ≥50% predicted at visit 1.
5. DLCO (corrected for hemoglobin) ≥30% predicted at visit 1.
6. Either:

   1. On a stable dose of licensed IPF therapy for at least 8 weeks prior to visit 1 and expected to remain on this background treatment after randomization. Due to the risk of DDIs, concomitant treatment with pirfenidone is not allowed in this trial.
   2. Not currently receiving treatment for IPF with a licensed therapy for any reason, including prior intolerance, non-responsiveness, ineligibility, lack of access or voluntarily decline. Any such previous treatment must have been discontinued >8 weeks prior to visit 1.
7. Anticipated life expectancy of at least 12 months at visit 1 and not anticipated to require a lung transplant during the trial period (being on a transplant list does not exclude a participant from the trial).
8. Contraceptive use by women of childbearing potential (WOCBP) which is highly effective and consistent with local regulations regarding the methods of contraception for those participating in clinical trials.

   For UK and countries within the EU: Male participants, if heterosexually active with a female partner of childbearing potential, or a pregnant or breastfeeding partner, must agree to use barrier contraception (male condom) and abstain from sperm donation for the duration of the treatment period and for at least 2 weeks after the last dose of the trial drug.
9. Written informed consent, consistent with ICH-GCP and local laws, obtained before the initiation of any trial-related procedure.

Exclusion Criteria

Participants are excluded from the trial if any of the following criteria apply:

1. Concurrent serious medical condition that in the opinion of the investigator constitutes a risk or a contraindication for participation in the trial or that could interfere with the trial objectives, conduct or evaluation, including active or suspected malignancy or history of malignancy within 5 years prior to visit 1, except appropriately treated basal cell carcinoma of the skin, fully resected and cured squamous cell carcinoma of the skin, "under surveillance" prostate cancer or in situ carcinoma of uterine cervix.
2. Airways obstruction with a pre-bronchodilator forced expiratory volume in one second (FEV1)/FVC ratio <0.7 at visit 1.
3. Lower respiratory tract infection requiring antibiotics and not fully recovered according to investigator judgement within 4 weeks prior to visit 2.
4. Confirmed infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) requiring hospitalization and not fully recovered according to investigator judgement within 4 weeks prior to visit 2.
5. Known impaired hepatic function or clinically significant liver disease (Child-Pugh B or C hepatic impairment), or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) or total bilirubin >1.5 times ULN at visit 1.
6. Severe renal impairment (i.e., estimated glomerular filtration rate (eGFR) ≤35 ml/min/1.73 m2 at visit 1 according to Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).
7. Prolonged QTcF (QT interval with Fridericia's correction) (>450 ms), AV-block II or III, uncontrolled arrhythmia, or other clinically significant abnormality in the resting ECG at visit 1, as judged by the investigator. Patients with implantable cardiovascular devices (e.g. pacemaker) affecting the QT interval time may be enrolled in the trial based upon investigator judgement, following cardiologist consultation if deemed necessary, and only after discussion with the medical monitor.
8. Heart failure NYHA Class IV, acutely decompensated right heart failure, PH with syncopal episode, confirmed myocardial infarction, unstable angina or uncontrolled hypertension, within 6 months prior to visit 1.
9. Known hypersensitivity or intolerance to buloxibutid or to any other components of the test product, including excipients.
10. Pregnant or breast-feeding female participants.
11. Acute IPF exacerbation within 3 months prior to visit 1 and/or during the screening period, as defined by Collard et al., 2016:

    1. Acute worsening or development of dyspnea typically <1 month duration.
    2. Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia pattern (if no previous computed tomography is available, the qualifier "new" can be dropped).
    3. Deterioration not fully explained by cardiac failure or fluid overload.
12. Inability to generate a spirometry test at visit 1 meeting the standards of the ATS/ERS 2019 guideline (Graham et al., 2019).
13. Treatment with pirfenidone within 8 weeks prior to visit 1 or anticipated need for pirfenidone during participation in the trial.

More exclusion criteria may apply.

Trial website: www.aspire-ipf.com

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of buloxibutid compared to placebo in participants with IPF as assessed by FVC | week 52
  • Absolute change from baseline in FVC (mL) at week 52

SECONDARY OUTCOMES:
To further evaluate the effects of buloxibutid on disease progression, respiratory-related hospitalization or death compared to placebo in participants with IPF | week 52
  • A composite of the proportion of patients with an absolute FVC percent predicted (FVCpp) decrease from baseline of ≥10%; a respiratory-related hospitalization, or death, up to week 52

CONTACTS AND LOCATIONS:
Locations (115):
- United States (29):
  - UAB Hospital, School of Medicine/Lung Health Center, Birmingham, Alabama
  - Keck Medicine of University of Southern California, Los Angeles, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - UC Davis Health System, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Paradigm Clinical Research, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida Health (UF Health), Gainesville, Florida
  - Clinical Research Specialists, Kissimmee, Florida
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Endeavor Health - Evanston Hospital, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Pulmonary & Critical Care Medicine, Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Renown Clinical Research, Reno, Nevada
  - University of New Mexico, Health Sciences Center, Albuquerque, New Mexico
  - Stony Brook University, Stony Brook, New York
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Cleveland Clinic - Cleveland, Department of Pulmonary Medicine, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Summit Health - Bend, Bend, Oregon
  - Oregon Clinic, Pulmonary, Critical Care & Sleep Medicine East, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Low Country Lung and Critical Care, North Charleston, South Carolina
  - StatCare - Bearden, Knoxville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - University of Utah, Health Sciences Center, Salt Lake City, Utah
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Argentina (11):
  - Research Institute of Respiratory Diseases, San Miguel de Tucumán, Tucumán Province
  - CEMER Medical Center for Respiratory Diseases, Buenos Aires
  - Belgrano Clinical Research Center, Buenos Aires
  - CINME - Metabolic Research Center, Buenos Aires
  - Medical Center Dra. De Salvo, Buenos Aires
  - IMER Respiratory Medicine Institute, Córdoba
  - Breathe Comprehensive Clinical Health, Godoy Cruz
  - Emphysema Foundation, Pneumology, Mar del Plata
  - Vistalba Health Center, Mendoza
  - InnovaCiencia, Rosario
  - Ibamedica, Santa Fe
- Australia (9):
  - Lung Research Victoria, Footscray, Victoria
  - Flinders Medical Centre, Adelaide
  - The Prince Charles Hospital, Brisbane
  - Concord Repatriation General Hospital, Department of Respiratory Medicine, Concord
  - St Vincent's Hospital, Sydney Ltd., Darlinghurst
  - Townsville University Hospital, Douglas
  - Austin Hospital, Heidelberg
  - Royal Prince Alfred Hospital, Sydney
  - The Queen Elizabeth Hospital, Woodville
- Austria (3):
  - Kepler University Hospital GmbH, Department of Pulmonology, Linz, Upper Austria
  - Salzburg Regional Hospital, Department of Pneumology/Respiratory Medicine, Salzburg
  - Hospital Penzing, Department of Respiratory and lung diseases, Vienna
- Belgium (4):
  - Erasme Hospital, Brussels
  - University Hospitals Saint-Luc, Brussels
  - University Hospital Center Sart-Tilman, Liège
  - UCL Mont-Godinne University Hospitals, Yvoir
- Canada (4):
  - Kelowna Respiratory & Allergy Clinic, Kelowna, British Columbia
  - Laval Hospital, Laval, Quebec
  - Pierre-Le Gardeur, Terrebonne, Quebec
  - Diex Research Trois-Riviere Inc., Trois-Rivières, Quebec
- Germany (7):
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital Heidelberg, Clinic of Thoracic Medicine Heidelberg GmbH, Heidelberg, Baden-Wurttemberg
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - Immenhausen Lung Hospital, Immenhausen, Hesse
  - Hannover Medical School, Center for Internal Medicine, Hanover, Lower Saxony
  - RuhrlandClinic - Lung Center, Essen, North Rhine-Westphalia
  - Vivantes Hospital Neukoelln, Berlin
- Greece (8):
  - University General Hospital of Heraklion, Pneumonology Clinic, Heraklion, Crete
  - "Sotiria" Chest Diseases Hospital of Athens, Athens
  - General Hospital of Chest Diseases "Sotiria" 5th Pulmonology Department, Athens
  - University General Hospital "Attikon", 2nd Pulmonary Department, Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
  - General Hospital of Thessaloniki "G. Papanikolaou", University Department of Pulmonology, Thessaloniki
- Italy (6):
  - IRCCS Policlinic Hospital San Martino, Genoa, Liguria
  - University Hospital - Ospedali Riuniti Umberto I - GM Lancisi - G Salesi of Ancona, Ancona
  - Local Healthcare Company Papa Giovanni XXIII (ASST Papa Giovanni XXIII), Bergamo
  - San Gerardo of Tintori IRCCS Foundation, Monza
  - Foundation PTV - Polyclinic Tor Vergata, Roma
  - University Hospital City of Health and Science of Turin - Hospital Molinette, Turin
- Mexico (4):
  - National Institute of Respiratory Diseases Ismael Cosio Villegas (INER), Mexico City, Mexico City
  - Dr. Jose Eleuterio Gonzalez Monterrey University Hospital, Monterrey, Nuevo León
  - Integral Health Medical Unit, San Nicolás de los Garza, Nuevo León
  - Oaxaca Site Management Organization S.C - (Osmo), Oaxaca City
- Poland (5):
  - MICS Medical Centre Bydgoszcz, Bydgoszcz
  - VITAMED Galaj i Cichomski General Partnership, Bydgoszcz
  - Norbert Barlicki University Clinical Hospital in Lodz Departament of Pneumology and Allergy, Lodz
  - Twoja Przychodnia Medical Centre of Nowa Sol, Nowa Sól
  - Allergology- Pulmunology Outpatient Clinic Alergopneuma, Pulmonology Outpatient Clinic, Świdnik
- South Korea (11):
  - Soon Chun Hyang Central Medical Center, Bucheon-si
  - The Catholic University Of Korea Bucheon St. Mary's Hospital, Bucheon-si
  - InJe University Busan Paik Hospital, Busan
  - InJe University Haeundae Paik Hospital, Busan
  - Hanyang University - Myongji Hospital, Goyang-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (7):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Devon and Exeter Hospital, Exeter
  - Homerton University Hospital, London
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- See also: Trial webpage — http://aspire-ipf.com